CLINICAL TRIAL: NCT02011646
Title: Testing a Healthy Weight Intervention in Adolescents
Brief Title: Healthy Body Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI changed institutions
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GCO 13-0765
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Obesity
Keywords: diet; body weight; eating; eating disorder; exercise
MeSH Terms: conditions — Obesity; Body Weight; Feeding and Eating Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Weight (Experimental): intervention four times per week and consist of approximately 10 participants.
  Interventions: Behavioral: Healthy Weight
- Controlled Intervention (Active Comparator): Participants will be given a copy of the DVD. They will also be given the choice to stream it free on the web.
  Interventions: Behavioral: Controlled Intervention

INTERVENTIONS:
Behavioral: Healthy Weight — The PI will train 4 group leaders to deliver the intervention. Groups will be offered four times per week and consist of approximately 10 participants. Each group will be led by 2 group leaders and each group leader will lead two sessions per week during the 2.5 mo intervention period. Group leaders will digitally video-record all sessions of the first two groups they deliver so the PI can provide supervision and rate fidelity and competence for a random selection of 6 of these 12 sessions. Group leaders will transmit the video recordings via an encrypted, secure internet connection to Dr. Ochner (who was trained by Dr. Eric Stice, the creator of the intervention) within 3 d for supervision, and competence and fidelity assessments.
  Arms: Healthy Weight
Behavioral: Controlled Intervention — "The Weight of the World" is a 51 min documentary focusing on the topics of obesity and healthy living. Via information presented by medical professionals and lifestyle experts, this film delves into issues related to preventing and combating obesity. Major topics include the importance of healthy eating and exercise behaviors and the changes that can be made by communities to reshape our lifestyles. Participants will be given a copy of the DVD. They will also be given the choice to stream it free on the web.
  Arms: Controlled Intervention

SUMMARY:
Few obesity prevention programs have produced weight gain prevention effects that persist over long-term follow-up and those that have are extremely lengthy, averaging 52 hr in duration, making implementation difficult and costly. The 2010 US Preventative Services Task Force (USPSTF) recommendations for treating child & adolescent obesity state that programs should have ≥ 25 hr of comprehensive treatment including dietary, physical activity and behavioral counseling, and that programs with < 25 hr usually do not produce improvements. The implication is that, if centers cannot provide this level of service (as most cannot), it is not worth providing any kind of treatment at all. In extreme exception to this, an intensive 3-hr non-restrictive obesity prevention program involving participant-driven healthy lifestyle improvement plans designed to bring caloric intake and output into balance (Healthy Weight) has been found to significantly reduce increases in BMI and obesity onset relative to alternative interventions and assessment-only controls through 3-yr follow-up. We propose to test an extended 6-hr version of the Healthy Weight intervention in a sample of primarily low SES, minority adolescents and young adults who are overweight and report body dissatisfaction and subthreshold eating disorder symptoms, as these are prevalent risk factors for obesity. We will test the hypothesis that participants assigned to the Healthy Weight vs. control intervention will have significantly lower BMI and % body fat during follow-up. Secondary outcomes will include body dissatisfaction, depressive symptoms, and eating disorder symptoms. 300 adolescents and young adults at high risk for future weight gain by virtue of their age, BMI percentile, body dissatisfaction and eating disorder symptomatology will be randomized to Healthy Weight or weight control educational video. Participants will complete assessments of BMI, body composition, potential mediators, and other outcomes at pretest, posttest and 6--mo follow-ups (in yr 1). Thus, to refute the USPSTF recommendations statement, we propose to show that a 6-hr intervention led by graduate students can produce significant reductions in risk for both obesity and eating disorders, suggesting this inexpensive and brief intervention could and should be rolled out nationwide.

Primary Aim: To test the hypothesis that Healthy Weight will significantly reduce increases in BMI, % body fat, and risk for onset of obesity during follow-up.

Secondary Aim: To test the hypothesis that Healthy Weight will significantly reduce body dissatisfaction, depressive symptoms, and eating disorder symptoms.

NOTE: THIS STUDY IS ONLY OPEN TO PATIENTS AT THE MOUNT SINAI ADOLESCENT HEALTH CENTER

DETAILED DESCRIPTION:
Obesity is associated with increased risk of mortality, atherosclerotic cerebrovascular disease, coronary heart disease, colorectal cancer and death from all causes (Flegal et al., 2005), is credited with over 111,000 deaths annually in the US (Flegal et al., 2005), shortens the lifespan by 5-20 years (Fontaine et al., 2003) and results in $150 billion in annual health-related expenditures (Finkelstein et al., 2009). Despite alarming increases in both adult and childhood obesity in recent decades, obesity rates in adolescents have grown at an even faster rate (Ogden et al., 2012; NCHS, 2012). Adolescent obesity has more than tripled in the past 30 years and continues to rise (Ogden et al., 2012; NCHS, 2012). Obese adolescents are more likely to have high cholesterol and high blood pressure, prediabetes, bone/joint problems, sleep apnea, and social and psychological problems such as stigmatization and poor self-esteem (DHHS, 2010; CDC, 2011). Unfortunately, virtually all obesity treatments result in only transient weight loss (Turk et al., 2009). Evidence suggests that it is nearly impossible for individuals to maintain behavioral weight losses once they have been obese for an extended period of time (Ochner et al., 2013). Although bariatric surgery can result in more persistent weight loss, this invasive procedure is contraindicated for numerous individuals, particularly children (Martin et al., 2010). Thus, a pressing public health priority is to develop simple and effective obesity prevention programs.

In 2010, the U.S. Preventive Services Task Force (USPSTF) issued recommendations for screening and treating childhood and adolescent obesity. They endorsed comprehensive moderate-to high intensity programs including counseling for weight loss, healthy diet, and physical activity as well as instruction and support for the use of behavioral management techniques including self-monitoring, stimulus control, eating management, contingency management, and cognitive behavioral therapy techniques. The USPSTF further defined moderate- to high-intensity programs as > 25 hr of contact and states that "such interventions would not be feasible for implementation in a primary care setting." (USPSTF, 2010, p. 365). Further, they assert that less intensive (< 25 contact hours) programs do not produce significant improvements. "Low-intensity interventions, defined as < 25 contact hours over a 6-month period, did not result in significant improvement in weight status" (USPSTF, 2010, p. 364). The implication is that, since most centers cannot provide this level of service, it is not worthwhile for adolescent health centers to provide any kind of obesity intervention at all. According to the USPSTF's website, "its recommendations are considered the gold standard for clinical preventive services." Such recommendations could discourage the testing and implementation of brief interventions designed to prevent obesity. Thus, to refute USPSTF statement, we propose to show that a 6-hr intervention led by graduate students can produce significant reductions in risk for both obesity and eating disorders, suggesting that this brief and inexpensive intervention could and should be rolled out nationwide.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 12 years old
* Body image concerns
* Sub-threshold Eating disorder symptomatology
* Overweight but not obese (BMI between the 85th and 95th percentile for children/adolescents and BMI between 25 and 30 kg/m2 for adults 21-24)
* Be able to commit to weekly 1-hour sessions for six weeks and 3 separate assessment visits to the MSAHC

Exclusion Criteria:

* Current eating disorder (anorexia nervosa, bulimia nervosa or binge eating disorder)
* absence of body image concerns
* normal or obese body weight (< 85th or ≥ 95th BMI percentile)

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2013-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | baseline
  Height will be measured to the nearest millimeter using a direct reading stadiometer. Weight will be assessed to the nearest 0.1 kg using a digital scale (Tanita TBF-300A) with participants wearing light clothing without shoes or coats.
Body Mass Index (BMI) | at 5 min post intervention
  Height will be measured to the nearest millimeter using a direct reading stadiometer. Weight will be assessed to the nearest 0.1 kg using a digital scale (Tanita TBF-300A) with participants wearing light clothing without shoes or coats.
Body Mass Index (BMI) | 6 month follow-up
  Height will be measured to the nearest millimeter using a direct reading stadiometer. Weight will be assessed to the nearest 0.1 kg using a digital scale (Tanita TBF-300A) with participants wearing light clothing without shoes or coats.
Body Fat | baseline
  Body Fat - We will use bioelectrical impedance analysis (BIA) using the Tanita TBF-300A Body Composition Analyzer to assess % body fat to maximize our sensitivity to predict increases in body fat and obesity onset. Two measures will be averaged.
Body Fat | at 5 min post intervention
  Body Fat - We will use bioelectrical impedance analysis (BIA) using the Tanita TBF-300A Body Composition Analyzer to assess % body fat to maximize our sensitivity to predict increases in body fat and obesity onset. Two measures will be averaged.
Body Fat | 6 month follow up
  Body Fat - We will use bioelectrical impedance analysis (BIA) using the Tanita TBF-300A Body Composition Analyzer to assess % body fat to maximize our sensitivity to predict increases in body fat and obesity onset. Two measures will be averaged.

SECONDARY OUTCOMES:
Body Dissatisfaction | baseline
  an adapted form of the Satisfaction and Dissatisfaction with Body Parts Scale to assess body satisfaction (Berscheid et al., 1973). It asks respondents to rate their level of satisfaction with nine body parts on 6-point scales ranging from "extremely satisfied" to "extremely dissatisfied." This scale has shown excellent internal consistency, temporal reliability, predictive validity for eating disorder symptom onset, and sensitivity to intervention effects (Stice et al., 2006; 2008; 2012).
Body Dissatisfaction | at 5 min post intervention
  an adapted form of the Satisfaction and Dissatisfaction with Body Parts Scale to assess body satisfaction (Berscheid et al., 1973). It asks respondents to rate their level of satisfaction with nine body parts on 6-point scales ranging from "extremely satisfied" to "extremely dissatisfied." This scale has shown excellent internal consistency, temporal reliability, predictive validity for eating disorder symptom onset, and sensitivity to intervention effects (Stice et al., 2006; 2008; 2012).
Body Dissatisfaction | at 6 months follow up
  an adapted form of the Satisfaction and Dissatisfaction with Body Parts Scale to assess body satisfaction (Berscheid et al., 1973). It asks respondents to rate their level of satisfaction with nine body parts on 6-point scales ranging from "extremely satisfied" to "extremely dissatisfied." This scale has shown excellent internal consistency, temporal reliability, predictive validity for eating disorder symptom onset, and sensitivity to intervention effects (Stice et al., 2006; 2008; 2012).
Eating Disorders | baseline
Eating Disorders | at 5 min post intervention
Eating Disorders | at 6 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ochner, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States